CLINICAL TRIAL: NCT02007460
Title: The Influence of High Impact Exercise on Musculoskeletal Health in Older Men
Acronym: Hiphop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: University Hospitals Leicester NHS Trust, UK (Unknown); University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Katherine Brooke-Wavell, Senior Lecturer in Human Biology, Loughborough University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: R10-P1
Record Dates: First submitted 2013-11-27; First posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Bone Strength; Neuromuscular Function
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise leg (Experimental)
  Interventions: Behavioral: Exercise
- Control leg (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — multidirectional unilateral hopping exercise
  Arms: Exercise leg

SUMMARY:
Osteoporotic fractures are an extremely common and serious public health issue which contribute substantially to pain, impaired mobility and morbidity in the elderly. Declines in bone strength combined with an increase risk of falls (associated with decline in muscular function with age) are the main determinants of fracture risk. Exercise that is novel and involves impact loading has the potential to improve bone strength and neuromuscular function (strength, power and balance). It is thus imperative to evaluate potential benefits of exercise in older people. The musculoskeletal responses to exercise may also be influenced by vitamin D status. It is the purpose of this study to consider the influence of a one year unilateral (one limb) high impact exercise programme on musculoskeletal health, specifically bone structure, muscle strength and power in older caucasian men. It is also the purpose of this study to determine whether this differs according to vitamin D status. The findings will reveal whether exercise can improve bone health and/or neuromuscular function, and whether improvements are dependent upon vitamin D status.

ELIGIBILITY:
Inclusion Criteria:

* Healthy community dwelling men of white european origin

Exclusion Criteria:

* BMI >30 kg/m2
* History of strength training or recently ( previous 12 months) doing moderate physical activity (weight bearing, high impact)
* Recent ( previous 12 months) or current medical or surgical problems likely to affect bone metabolism or provide contraindications to high impact exercise, balance or neuromuscular function
* Any previous or existing lower back or limb problems that could be exacerbated by undertaking high impact exercise
* Any history of diagnosed or symptomatic diseases likely to influence strength, power, bone or habitual activity (including osteomalacia or impaired liver/renal function and locomotor disease, hypertension) that influences bone or muscle or precludes exercise

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in femoral neck bone mineral density | baseline, 12 months

SECONDARY OUTCOMES:
Change in cortical bone mineral content | baseline, 12 months
Change in trabecular bone mineral content | baseline, 12 months
Change in ground reaction force during hopping | baseline, 6 months, 12 months
Change in electromyography of quadriceps during hopping | baseline, 6 months
Change in postural sway amplitude (mm) | baseline, 6 months
Change in leg press strength | baseline, 6 months
Change in maximal isometric knee extensor strength | baseline, 6 months
Change in tendon stiffness | baseline, 6 months

OTHER OUTCOMES:
Serum 25 hydroxy vitamin D | baseline
Change in body fat content | baseline, 12 months
change in energy intake (MJ/d) | baseline, 12 months
change in calcium intake | baseline, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Brooke-Wavell, PhD, Principal Investigator — Loughborough University; Winston Rennie, MBBS, Principal Investigator — University Hospitals Leicester NHS Trust; Jonathan Folland, PhD, Principal Investigator — Loughborough University; Greg Summers, MD, Principal Investigator — Derby University Hospitals Trust
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

REFERENCES:
- [Result] Allison SJ, Folland JP, Rennie WJ, Summers GD, Brooke-Wavell K. High impact exercise increased femoral neck bone mineral density in older men: a randomised unilateral intervention. Bone. 2013 Apr;53(2):321-8. doi: 10.1016/j.bone.2012.12.045. Epub 2013 Jan 3. PMID 23291565